CLINICAL TRIAL: NCT01321970
Title: Validation and Evaluation of Multimodal Imaging Combining Three-dimensional Ultrasound and Stress Myocardial Scintigraphy in the Diagnosis of Coronary Artery Disease
Brief Title: Validation/Evaluation of Multimodal Imaging Combining 3D Ultrasound and Stress Myocardial Scintigraphy in the Diagnosis of Coronary Artery Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Impossible to start to the study.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI/2009/VB-01
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2015-03

CONDITIONS: Coronary Artery Disease; Coronary Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Severe coronary artery disease (Other): Patients in this group have coronary artery disease with a stenosis of >70%.
  Interventions: Procedure: Stress ultrasound; Procedure: Scintigraphy; Procedure: Coronary angiography
- Coronary artery disease (Other): Patients in this group have coronary artery disease with stenosis < 70%.
  Interventions: Procedure: Stress ultrasound; Procedure: Scintigraphy; Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Stress ultrasound — Qualitative interpretation of the left ventricular wall motion abnormalities is performed in real time in the resting phase and during pharmacological stress. The translation of quantitative data is then performed for each of the 17 segments on a bulls-eye pattern identical to that of scintigraphy.
Procedure: Scintigraphy — Image acquisition is synchronized to the electrocardiogram. The tomographic sections are represented in the 3 directions of space, the analysis is also done on the classical representation in 17 segments. (Typically used in ultrasound perfusion scintigraphy or PET).
Procedure: Coronary angiography — Performed in interventional cardiology setting using a guide introduced through the radial or femoral artery. The injection of iodine allows opacification of coronary arteries and their visualization by fluoroscopy. The qualitative interpretation of the data is translated in terms of percentage of stenosis of the coronary artery. It is thus considered that the stenosis is significant at over 70% obstruction of the lumenal diameter. This interpretation is made for each of the three main coronary arteries and their tributaries:
  * Right coronary (proximal, middle and distal) and collateral (inter ventricular posterior ventricular posterior retro)
  * Inter ventricular anterior (proximal, middle and distal) and its tributaries (diagonal and septal)
  * Circumflex (proximal, middle and distal) and collateral (first and second marginal)

SUMMARY:
Our primary goal is to validate a new diagnostic tool for functional coronary artery stenosis that uses multimodal imaging (combining stress echocardiography and stress scintigraphy) in patients with known coronary chest pain.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has a documented coronaropathy
* The patient needs a new coronarography following symptoms indicating a change in his/her coronary disease state

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* Patients with arrhythmias, left bundle branch block on the electrocardiogram which would complicate the interpretation of examinations
* Unstable, acute coronary syndromes unstable needing emergency coronary angiography
* Patient with contraindication for conducting a stress test:
* poorly controlled hypertension
* pre-existing severe arrhythmia
* aortic stenosis
* and obstructive hypertrophic cardiomyopathy
* Patient has contraindication for atropine
* History of prostate adenoma
* Glaucoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The difference between AUCs for multimodal imaging and scintigraphy | 4 days

SECONDARY OUTCOMES:
The difference between AUCs for multimodal imaging and stress ultrasound | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Rubini, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France